CLINICAL TRIAL: NCT04170374
Title: Survey of Procedures and Resources for Initiating Treatment of HIV in Africa: The SPRINT Study in South Africa
Brief Title: Survey of Procedures and Resources for Initiating Treatment of HIV in Africa-South Africa
Acronym: SPRINT-SA
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University of Witwatersrand, South Africa (Other)
Responsible Party: Sponsor
Other Study IDs: H-39330; OPP1136158 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: HIV; Antiretroviral Therapy
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who initiated HIV treatment
  Interventions: Other: Routine medical record data collection
- Service providers at study facilities
  Interventions: Other: Interviews with service providers

INTERVENTIONS:
Other: Routine medical record data collection — The study will collect routine medical record data from the electronic medical record system, other electronic databases, and paper charts.
  Groups: Patients who initiated HIV treatment
Other: Interviews with service providers — Clinicians and lay staff will be interviewed regarding the ART initiation process.
  Groups: Service providers at study facilities

SUMMARY:
In its 2017 revision of the global guidelines for HIV care and treatment, the World Health Organization called for rapid or same-day initiation of antiretroviral treatment (ART) for eligible patients testing positive for HIV. The South African National Department of Health adopted this recommendation in October 2017. Neither organization provided detailed guidance, however, on how to implement the recommendation.

In sub-Saharan Africa, where most HIV patients are located, studies continue to document high losses of treatment-eligible patients from care before they receive their first dose of antiretroviral medications (ARVs). Among facility-level reasons for these losses are treatment initiation protocols that require multiple clinic visits and long waiting times before a patient who tests positive for HIV is dispensed an initial supply of medications. There is very little published evidence on the practical details of the process and the extent to which it varies by facility, setting, or country. Without a robust baseline evidence base, it is challenging to identify opportunities for making improvements. The SPRINT (Survey of Procedures and Resources for Initiating Treatment of HIV in Africa) study will begin to develop this evidence base. SPRINT will combine a facility-level description of the standard of care with a retrospective record review of patients who recently initiated ART at the study sites. Data will be collected from 12 clinics across 3 provinces in South Africa (KwaZuluNatal Province, Gauteng Province, and Limpopo Province). The survey will elicit detailed information about current procedures through structured interviews with clinic staff. The record review for a retrospective cohort of patients eligible for ART will estimate actual numbers of clinic visits, services provided, and duration of the steps for treatment initiation from start to finish. SPRINT is expected to identify differences in approaches to treatment initiation and potential opportunities for improvement.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* HIV-positive

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who became eligible for ART at a study facility between 1 January 2018 and 31 December 2018.
Sampling Method: Non-Probability Sample
Enrollment: 831 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Average numbers of visits required to start ART | Up to 6 months after treatment eligibility determined
  Number of health system interactions required between HIV diagnosis and first dispensing of ARVs
Time to ART initiation | Up to 6 months after treatment eligibility determined
  Average number of days required between HIV diagnosis and first dispensing

CONTACTS AND LOCATIONS:
Overall Officials: Sydney B Rosen, MPA, Principal Investigator — BU School of Public Health
Locations (1):
- Amy Huber, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huber A, Hirasen K, Brennan AT, Phiri B, Tcherini T, Mulenga L, Haimbe P, Shakwelele H, Nyirenda R, Wilson Matola B, Gunda A, Rosen S. Uptake of same-day initiation of HIV treatment in Malawi, South Africa, and Zambia as reported in routinely collected data: the SPRINT retrospective cohort study. Gates Open Res. 2023 May 2;7:42. doi: 10.12688/gatesopenres.14424.2. eCollection 2023. PMID 37153118